CLINICAL TRIAL: NCT04447365
Title: The Correlation Between Gut Microbiome-host Interaction and Ventricular Arrhythmias.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: North Florida Foundation for Research and Education (Other)
Responsible Party: Sponsor
Other Study IDs: 202001134
Record Dates: First submitted 2020-06-22; First posted 2020-06-25 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Gut Microbiome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: 10 patients who have had no device-monitored for ventricular tachycardia/ ventricular fibrillation the 3 months prior to recruitment will comprise a group of controls
  Interventions: Diagnostic Test: device interrogation
- high burden of ventricular arrhythmias: 20 patients will comprise a group of patients with high burden of ventricular arrhythmias, defined as patients with at least one sustained episode of VT/VF requiring ICD therapies in the 3 months preceding study enrollment.
  Interventions: Diagnostic Test: device interrogation

INTERVENTIONS:
Diagnostic Test: device interrogation — All patients will have a pre-existing ICD and a diagnosis of cardiomyopathy with left ventricular systolic function of 35% or less by echocardiogram done within 3 years of the time of enrollment.

SUMMARY:
This study will enroll 30 subjects recruited from the electrophysiology device clinic at the VA medical center. All patients will have a pre-existing implantable cardioverter defibrillator and a diagnosis of cardiomyopathy with left ventricular systolic function of 35% or less by echocardiogram done within 3 years of the time of enrollment. 10 patients who have had no device-monitored ventricular fibrillation/ ventricular tachycardia for the 3 months prior to recruitment will comprise a group of controls. 20 patients will comprise a group of patients with high burden of ventricular arrhythmias, defined as patients with at least one sustained episode of ventricular tachycardia/ ventricular fibrillation requiring implantable cardioverter-defibrillator therapies in the 3 months preceding study enrollment. This information will be obtained from device interrogation at the time of recruitment. Patients will provide a fecal sample for analysis at the time of enrollment.

DETAILED DESCRIPTION:
The investigators will recruit patient from the VA pacemaker/ implantable cardioverter defibrillator clinic. Patients with ICDs will be identified before scheduled clinical visit. Patients whose ICDs on remote monitoring show evidence of VT/VF and who are being admitted to the VA medical center for expedited inpatient work up and treatment will also be offered enrollment in the study. Patients will be approached and educated about the study rationale and their involvement. Patients will be consented for participation in the study after their approval. Patients will be educated about donating fecal samples. Patients will be given fecal sampling kits to collect and subsequently mail in those samples to the University of Florida physiology laboratory where there will be processed in a HIPAA compliant way. These samples will be subjected to laboratory analysis which will be outsourced. Fecal samples will be analyzed by shotgun metagenomics to characterize the taxonomy of the gut flora and compare the taxonomic and physiologic differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* • age >18 years-old

  * competent and willing to provide consent
  * presence of implantable cardioverter-defibrillator
  * diagnosis of cardiomyopathy
  * left ventricular ejection fraction of 35% or less as assessed by echocardiogram within 3 years prior to enrollment

Inclusion criteria for control group:

• no VT/VF on device interrogation for a period of at least 3 months preceding study enrollment

Inclusion criteria for high ventricular arrhythmia burden group:

• at least one episode of sustained VT/VF or VT/VF requiring ICD therapies within the preceding 3 months as assessed on device interrogation at the time of study enrollment

Exclusion Criteria:

* • currently pregnant or have been pregnant in the last 6 months

  * antibiotic treatment within 5 months of study enrollment (i.e. antibiotic therapy in the two months prior to the 3-month period of analysis for VT/VF)
  * chronic use of medications/supplements that can potentially affect gut microbiota (i.e. probiotics, anti-inflammatory agents, glucocorticoids, other immune modulating medications, antacids or proton pump inhibitors)
  * history of intestinal surgery, inflammatory bowel disease, celiac disease, lactose intolerance, chronic pancreatitis, or other malabsorption disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Differences in gut microbiome in patients prone to clinically significant ventricular arrhythmias compared with matched controls with no ventricular arrhythmias. Evaluate potential clinical implications of the gut microbiome as it relates to ventricular arrhythmia burden and severity. Patients with an ICD and underlying cardiomyopathy to analyze fecal samples. The patients with high burden will be re-tested after undergoing a period of treatment for their arrhythmias and demonstrating a 3 month period wherein there are no recurrent device therapies. Fecal analysis of the groups will be compared.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
high burden arrhythmias | initially to 3 months
  : To identify specific gut microbiome characteristics of patients who are prone to clinically significant or high burden of ventricular arrhythmias
low burden arrhythmias | initially to 3 months
  To identify specific gut microbiome characteristics of patients with similar conventional risk factors and low burden of ventricular arrhythmias.
gut microbiome composition | 3 months
  : To examine changes that occur in the gut microbiome composition after treatment of ventricular arrhythmias.

CONTACTS AND LOCATIONS:
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No